CLINICAL TRIAL: NCT01793038
Title: Clomiphene Citrate Plus HPuFSH Versus Letrozole Plus HPuFSH in Clomid Resistant Infertile PCOS Women
Brief Title: Clomiphene Citrate Plus uFSH Versus Aromatase Inhibitor Plus uFSH in Clomiphene Resistant Infertile PCOS Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura Integrated Fertility Center (Other)
Responsible Party: Principal Investigator, Mohamad Elsaid Ghanem, Dr, Mansoura Integrated Fertility Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mific-3
Record Dates: First submitted 2013-02-10; First posted 2013-02-15 (Estimated); Last update posted 2013-03-06 (Estimated); Status verified 2013-03

CONDITIONS: Polycystic Ovary Syndrome; Infertility
Keywords: PCOS; clomiphene citrate resistant PCOS; Aromatase inhibitors
MeSH Terms: conditions — Polycystic Ovary Syndrome; Infertility | interventions — Aromatase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CC-plus uFSH (Active Comparator): clomiphene citrate 50 mg tablets twice/day for cycle days 3-7 plus daily IM injection of 37.5 IU HP uFSH for days 3-12
  Interventions: Drug: clomiphene citrate-uFSH arm
- Aromataze inhibitor plus uFSH (Experimental): Aromataze inhibitor (litrezole )2.5 mg twice daily for cycle days 3-7 plus daily IM injection of uFSH 37.5 IU for cycle days 3-12
  Interventions: Drug: Aromatase inhibitor (litrezole) plus uFSH arm

INTERVENTIONS:
Drug: Aromatase inhibitor (litrezole) plus uFSH arm — literozole tablets 5 mg /day for days 3-7 plus intramuscular injections of uFSH 37.5 IU/day for days 3-12
  Arms: Aromataze inhibitor plus uFSH
Drug: clomiphene citrate-uFSH arm — clomiphene citrate 50 mg tablets twice /day for 5 days plus 37.5 IU uFSH IM injections daily for 10 days
  Arms: CC-plus uFSH

SUMMARY:
Polycystic ovarian syndrome (PCOS) is a condition characterized by infertility, infrequent periods and amenorrhea or irregular bleeding plus anovulatory infertility. Clomid is the standard first drug of treatment for ovulation induction. Ovulation and conception will occur in approximately 75 and 30 percent of cases respectively. Cases not ovulating in response to doses of clomid up to 150 mg/day are known as clomid resistant PCOS.

DETAILED DESCRIPTION:
To test whether CC co- treatment with chronic low dose HP uFSH versus lirizole plus chronic low dose HP uFSH in CC resistant PCOS will yield comparable results in terms of, ovulation rate, lower follicle number, lower HP uFSH dose, better outcome in terms of pregnancy rates, better cost-effectiveness ratio, lower multiple pregnancy rates, lower cycle cancellation.

ELIGIBILITY:
Inclusion Criteria:

* CC resistant PCOS
* Infertile
* Females
* Age 18-38

Exclusion Criteria:

* Hyperprolactinaemia
* Cushing syndrome
* Adult onset adrenal hyperplasia
* Age > 38
* Other infertility factors in the couple than PCOS: male factor,tubal factor,edometriosis

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2013-03; Primary Completion 2014-06 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
ovulation rate | 30 days
  percentage of ovulatory cycles per started and per completed cycles

SECONDARY OUTCOMES:
endometrial thickness | 4 weeks
  endmetrial thickness at time of ovulation triggering
ongoing cycle pregnancy rate | 16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura Integrated fertility center, Al Mansurah, Dekahlia, Egypt

REFERENCES:
- [Background] Abdellah MS. Reproductive outcome after letrozole versus laparoscopic ovarian drilling for clomiphene-resistant polycystic ovary syndrome. Int J Gynaecol Obstet. 2011 Jun;113(3):218-21. doi: 10.1016/j.ijgo.2010.11.026. Epub 2011 Apr 1. PMID 21457973
- [Background] Palomba S, Falbo A, Zullo F. Management strategies for ovulation induction in women with polycystic ovary syndrome and known clomifene citrate resistance. Curr Opin Obstet Gynecol. 2009 Dec;21(6):465-73. doi: 10.1097/GCO.0b013e328332d188. PMID 19809318